CLINICAL TRIAL: NCT06645119
Title: Acute Effects of Protein Ingestion on Bone Turnover Biomarkers in Endurance Runners
Brief Title: Protein Ingestion on BMM Response in Endurance Runners
Acronym: BonePRO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Jenna Gibbs, Dr. Jenna Gibbs, Assistant Professor, McGill University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PRO-ENDO BONE
Record Dates: First submitted 2023-11-30; First posted 2024-10-16 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Dietary Proteins; Acute Exercise; Bone Diseases, Metabolic
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whey Protein Beverage (Experimental): Chocolate flavoured whey protein supplement as a post-exercise recovery beverage. One beverage post-exercise. Dose based on participant body weight.
  Interventions: Dietary Supplement: Whey Protein Supplement
- Control Beverage (Sham Comparator): Water beverage with calorie-free chocolate syrup as a post-exercise recovery beverage. Isovolumetric.
  Interventions: Dietary Supplement: Whey Protein Supplement

INTERVENTIONS:
Dietary Supplement: Whey Protein Supplement — Examining the independent effect of post-exercise dietary protein ingestion on bone metabolic markers.

SUMMARY:
The goal of this clinical trial is to investigate the effects of protein ingestion post-exercise on bone turnover markers. The main questions it aims to answer is:

Does protein ingestion independently influence the bone metabolic response to exercise in endurance runners?

We will compare dietary protein to a placebo (water) to detect changes in bone turnover markers.

Participants will:

In a within-subject design, participants will perform an exhaustive run and take either protein or placebo immediately post-exercise.

Track physical activity and diet before each arm of the intervention and during the washout period.

DETAILED DESCRIPTION:
Endurance athletes are at increased risk for bone loss and injury due to high-volume training, muscle weakness, and elevated nutritional demand. Dietary practices influence short- and long-term bone health and nutrition supplementation post-exercise may improve the short-term response of bone to exercise and benefit musculoskeletal recovery. However, we have a limited understanding of which dietary practices are most beneficial to optimize bone health in athletic populations. Protein supplementation has long been recommended for muscle adaptation and athletic performance but its potential for bone health has not been thoroughly investigated in endurance athletes. The purpose of this study is to is to investigate the acute independent effects of dietary protein ingestion on bone metabolism in healthy adults aged 18-35 years participating in high-volume endurance running.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years of age
* Healthy-range body mass index (BMI) (18.5-24.9 kg/m2)
* Competitive runner for at least one season (minimum 40 km/week for the past 6-months)
* Can read, speak, and understand French and/or English

Exclusion Criteria:

* Disease or medication known to affect bone metabolism
* Disease (e.g., uncontrolled thyroid disease, malabsorptive or inflammatory disorder, metabolic bone disease)
* Medication (e.g., hormonal contraceptives the past 3 months, glucocorticoids, anti-hypertensive drugs, anti-epileptic drugs, osteoporosis therapy)
* Orthopedic or musculoskeletal injury/disease that limits the capacity to exercise
* Current smoker or tobacco user
* Current diagnosis of an eating disorder
* Female participants with self-reported or diagnosed:
* Hypothalamic amenorrhea
* Polycystic ovarian syndrome
* Hyperprolactinemia
* Primary ovarian insufficiency
* Pregnant or breastfeeding
* Donated blood within the past two months

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Beta-C-terminal telopeptide | Up to 24 hours
  Bone resorption marker
Procollagen 1 Intact N-Terminal Propeptide | Up to 24 hours
  Bone formation marker

SECONDARY OUTCOMES:
Insulin-like growth factor 1 | Up to 24 hours
  Hormone involved in bone metabolism
Sclerostin | Up to 24 hours
  Bone turnover maker related to inflammatory response
OPG | Up to 24 hours
  Marker related to bone metabolic response
RANK/RANKL | Up to 24 hours
  Markers related to bone metabolic response
IL-6 | Up to 24 hours
  Marker related to bone metabolic response

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Gibbs, PhD, Principal Investigator — McGill University
Locations (1):
- McGillU, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferreira S, Gardy S, Linardatos J, Churchward-Venne T, Josse A, Correa J, Gibbs J. Acute effects of dietary whey protein supplementation after endurance exercise on serum osteokine and inflammatory cytokine concentrations in endurance runners. Appl Physiol Nutr Metab. 2026 Jan 1;51:1-15. doi: 10.1139/apnm-2025-0346. PMID 41506728